CLINICAL TRIAL: NCT03991260
Title: SPECT Imaging of HER2 Expression in Breast Cancer Using Technetium-99m-labelled ADAPT6
Brief Title: 99mTc-ADAPT6-based HER2 Imaging in Breast Cancer
Acronym: 99mTc-ADAPT6
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: KTH Royal Institute of Technology (Other); Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 99mTc-ADAPT6; 99mTc-ADAPT6 [TomskNRMC] (Other: TomskNRMC)
Record Dates: First submitted 2019-06-06; First posted 2019-06-19 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: 99mTc-ADAPT6; Breast Cancer; HER2 expression
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, Emission-Computed, Single-Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The tested injected doses of 99mTc- ADAPT6 500 µg: At least five (5) evaluable subjects with HER2-positive status and at least three (3) subjects with HER2-negative status have to be enrolled in the study for each tested protein dose. The tested injected dose is 500 µg. Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Diagnostic Test: SPECT
- The tested injected doses of 99mTc- ADAPT6 1000 µg: At least five (5) evaluable subjects with HER2-positive status and at least three (3) subjects with HER2-negative status have to be enrolled in the study for each tested protein dose. The tested injected dose is 1000 µg. Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Diagnostic Test: SPECT

INTERVENTIONS:
Diagnostic Test: SPECT — One single injection of 99mTc- ADAPT6, followed by gamma camera imaging directly post-injection and after 2, 4 and 6 hours.

SUMMARY:
The study should evaluate distribution of 99mTc- ADAPT6 in patients with primary HER2-positive and HER2-negative breast cancer.

The primary objective are:

1. To assess distribution of 99mTc- ADAPT6 in normal tissues and in tumours over time;
2. To assess kinetics of 99mTc- ADAPT6 in blood;
3. To evaluate dosimetry of 99mTc- ADAPT6;
4. To obtain initial information concerning safety and tolerability of 99mTc- ADAPT6 after single intravenous injection:

The secondary objective is:

1.To compare the tumour imaging data with the concerning HER2 expression obtained by immunohistochemistry (IHC) or fluorescent in situ hybridisation (FISH) analysis of biopsy samples:

DETAILED DESCRIPTION:
Overall goal of the project: To determine HER2 expression level in primary breast cancer and possibly in axillary lymph node metastases before neoadjuvant trastuzumab therapy.

Phase I. Distribution of 99mTc-ADAPT6 in patients with primary breast cancer. The study should evaluate distribution of 99mTc- ADAPT6 in patients with primary HER2-positive and HER2-negative breast cancer.

The primary objective are:

1. To assess distribution of 99mTc- ADAPT6 in normal tissues and in tumours over time;
2. To assess kinetics of 99mTc- ADAPT6 in blood;
3. To evaluate dosimetry of 99mTc- ADAPT6;
4. To obtain initial information concerning safety and tolerability of 99mTc- ADAPT6 after single intravenous injection:

The secondary objective is:

1. To compare the tumour imaging data with the concerning HER2 expression obtained by immunohistochemistry (IHC) or fluorescent in situ hybridisation (FISH) analysis of biopsy samples:

Methodology:

Open-label, exploratory, single centre study. The subjects will receive a single injection of the labelled tracer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Diagnosis of primary breast cancer with possible lymph node metastases
3. Availability of results from HER2 status previously determined on material from the primary tumor, either

   1. HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive or
   2. HER2-negative, defined as a DAKO HercepTest™ score of 0 or 1+; or else if 2+ then FISH negative
4. Volumetrically quantifiable tumour lesions on CT or MRI, with at least one lesion > 1.0 cm in greatest diameter outside of the liver and kidneys
5. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 10^9/L
   * Haemoglobin: > 80 g/L
   * Platelets: > 50.0 x 10^9/L
   * ALT, ALP, AST: =< 5.0 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
6. A negative pregnancy test (serum beta-human chorionic gonadotropin, beta-HCG) at screening for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
7. Subject is capable to undergo the diagnostic investigations to be performed in the study

11. Informed consent

Exclusion Criteria:

1. Second, non-breast malignancy
2. Active current autoimmune disease or history of autoimmune disease
3. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
4. Known HIV positive or chronically active hepatitis B or C
5. Administration of other investigational medicinal product within 30 days of screening
6. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with primary HER2-positive and HER2-negative breast cancer.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
Gamma camera-based whole-body 99mTc-ADAPT6 uptake value (%) | 6 hours
  Whole-body 99mTc-ADAPT6 uptake coinciding with normal organs and tissues will be assessed using gamma camera and calculated as percentage (%) of the injected dose of the radiopharmaceutical
SPECT-based 99mTc-ADAPT6 uptake value in tumor lesions (kcounts) | 6 hours
  99mTc-ADAPT6 uptake coinciding with tumor lesions will be assessed using single-photon emission computed tomography and measured in kcounts
SPECT-based 99mTc-ADAPT6 background uptake value (kcounts) | 6 hours
  Focal uptake of 99mTc-ADAPT6 in the regions without pathological findings will be assessed with SPECT and measured in kcounts
Tumor-to-background ratio (SPECT) | 6 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-ADAPT6 uptake coinciding with tumor lesions (kcounts) will be divided by the value of 99mTc-ADAPT6 uptake coinciding with the regions without pathological findings (kcounts)

SECONDARY OUTCOMES:
Safety attributable to 99mTc-ADAPT6 injections (physical findings) | 24 hours
  The safety attributable to 99mTc-ADAPT6 injections will be evaluated based on the assessments of physical examination, vital signs, and ECG (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-ADAPT6 injections (laboratory tests) | 24 hours
  The safety attributable to 99mTc-ADAPT6 injections will be evaluated based on the blood and urine laboratory tests (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-ADAPT6 injections (incidence and severity of adverse events) | 24 hours
  The safety attributable to 99mTc-ADAPT6 injections will be evaluated based on the rate of adverse events (%)
Safety attributable to 99mTc-ADAPT6 injections (concomitant medication) | 24 hours
  The safety attributable to 99mTc-ADAPT6 injections will be evaluated based on the rate of administration of concomitant medication (%)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, MD, Prof., Principal Investigator — TomskNMRC
Locations (1):
- TomskNRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No